CLINICAL TRIAL: NCT06769997
Title: The Optizum Study: A Randomized, Blinded Single Center Study Evaluating the Optilume BPH Catheter System and the Rezum Water Vapor Therapy for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Evaluation of the Optilume BPH Catheter System and the Rezum Water Vapor Therapy in Treating Benign Prostatic Hyperplasia
Acronym: OptiZum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-12549
Record Dates: First submitted 2024-10-16; First posted 2025-01-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Lower Urinary Track Symptoms
Keywords: Benign Prostatic Hyperplasia; Lower Urinary Track Symptoms; BPH; LUTS; Optilume; Rezum
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Randomized study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Optilume® BPH Catheter System (Active Comparator)
  Interventions: Device: Optilume® BPH Catheter System
- Rezum Water Vapor Therapy (Active Comparator)
  Interventions: Device: Rezum Water Vapor Therapy

INTERVENTIONS:
Device: Optilume® BPH Catheter System — The technology is based on a device/drug combination consisting of two catheters: the Optilume BPH Prostatic Pre-dilation Catheter which is a non-drug coated catheter used to start commissurotomy between the lateral lobes of the prostate and the Optilume BPH Prostatic Dilatation DCB Catheter which is a drug coated catheter used to complete the commissurotomy and transfers drug (paclitaxel) to the pre-dilated prostatic urethra and anterior commissure. Hence, the device applies a mechanical dilatation to open prostatic urethral lumen to increase urine flow, followed by the transfer of paclitaxel drug to inhibit cell proliferation and maintain this dilatation.
  Arms: Optilume® BPH Catheter System
Device: Rezum Water Vapor Therapy — The Rezum system is minimally invasive therapy for LUTS secondary to BPH. The system injects water vapor at 103°C generated by radiofrequency to create thermal energy via a transurethral approach. The vapor disperses through the tissue interstices within the treatment zone (transition zone). The injection of vapor last for approximatively 9 seconds and the number of injections depends on the prostate volume and length of the prostatic urethra.
  Arms: Rezum Water Vapor Therapy

SUMMARY:
Lower urinary symptoms (LUTS) affect older men and their frequency and severity increase with age. According to Berry et al., the histological diagnosis of benign prostatic hyperplasia (BPH) increases from 25% in the group age between 40 to 49 years to 80% in the group age between 70 to 79 years (1). However, this hyperplasia can lead to a bladder outlet obstruction (BOO) secondary to benign prostatic enlargement (BPE), causing storage and voiding symptoms, associated with a considerable impairment of the quality of life (2).

Surgical therapy of BPH has continuously evolved in recent years. The current gold standard for the endoscopic treatment of BPH is the transurethral resection of the prostate (TURP). Other innovative techniques were developed including Urolift, transurethral laser enucleation (holmium, thulium) and Aquablation therapy. One of the latest technologies for the management of BPH are Optilume BPH Catheter System (Optilume®, Urotronic Inc, Minneapolis, USA) and Rezum Water Vapor Therapy (Rezum System, Bostocn Scientific, Marlborough, MA).

The purpose of the present study is to compare between patient experience, symptom relief and functional improvement when using the Optilume BPH Catheter System (Optilume®, Urotronic Inc, Minneapolis, USA) and Rezum Water Vapor Therapy (Rezum System, Boston Scientific, Marlborough, MA).

DETAILED DESCRIPTION:
A- Background Lower urinary symptoms (LUTS) affect older men and their frequency and severity increase with age. According to Berry et al., the histological diagnosis of benign prostatic hyperplasia (BPH) increases from 25% in the group age between 40 to 49 years to 80% in the group age between 70 to 79 years. However, this hyperplasia can lead to a bladder outlet obstruction (BOO) secondary to benign prostatic enlargement (BPE), causing storage and voiding symptoms, associated with a considerable impairment of the quality of life.

Surgical therapy of BPH has continuously evolved in recent years. The current gold standard for the endoscopic treatment of BPH is the transurethral resection of the prostate (TURP). Other innovative techniques were developed including Urolift, transurethral laser enucleation (holmium, thulium) and Aquablation therapy. One of the latest technologies for the management of BPH are Optilume BPH Catheter System (Optilume®, Urotronic Inc, Minneapolis, USA) and Rezum Water Vapor Therapy (Rezum System, Bostocn Scientific, Marlborough, MA).

The Optilume BPH Catheter System was approved by the FDA in 2023. The technology is based on a device/drug combination consisting of two catheters: the Optilume BPH Prostatic Pre-dilation Catheter which is a non-drug coated catheter used to start commissurotomy between the lateral lobes of the prostate and the Optilume BPH Prostatic Dilatation DCB Catheter which is a drug coated catheter used to complete the commissurotomy and transfers drug (paclitaxel) to the pre-dilated prostatic urethra and anterior commissure. Hence, the device applies a mechanical dilatation to open prostatic urethral lumen to increase urine flow, followed by the transfer of paclitaxel drug to inhibit cell proliferation and maintain this dilatation.

The Rezum system is minimally invasive therapy for LUTS secondary to BPH. The system injects water vapor at 103°C generated by radiofrequency to create thermal energy via a transurethral approach. The vapor disperses through the tissue interstices within the treatment zone (transition zone). The injection of vapor last for approximatively 9 seconds and the number of injections depends on the prostate volume and length of the prostatic urethra.

The purpose of the present study is to compare between patient experience, symptom relief and functional improvement when using the Optilume BPH Catheter System (Optilume®, Urotronic Inc, Minneapolis, USA) and Rezum Water Vapor Therapy (Rezum System, Boston Scientific, Marlborough, MA).

B-Clinical experience

-Optilume® BPH Catheter System: The PINNACLE study was conducted by Kaplan et al. to evaluate the safety and efficacy of Optilume BPH when compared to a sham surgical procedure. The study was designed as a prospective, randomized, double-blinded, sham-controlled clinical trial. Eighteen participating centers in the United States and Canada recruited 148 patients over 50 years old with symptomatic BPH and a prostate size from 20 cc to 80 cc. Randomization assigned 100 patients to the Optilume BPH group and 48 patients to the sham procedure group. The primary endpoint was the comparison of the improvement in IPSS from baseline to 1 year in the Optilume BPH arm against 3 months in the sham arm. Other measurements included uroflowmetry, quality of life (QoL) and sexual function assessments. A blinded and independent clinical events committee prospectively collected data regarding adverse events (AE).

At one year, IPSS improved by 11.5 +/- 7.8 points in the Optilume BPH arm, which was significantly greater than the sham arm at 3 months (8.0 +/- 8.3). Additionally, QoL, sexual function, peak flow rate (Qmax) and post-void residual (PVR) significantly improved trough 1 year. Five serious adverse events probably related to the study device occurred including four hematuria and 1 urethral false passage. Other non-serious AEs included hematuria, urinary tract infection (UTI), dysuria, incontinence, bladder spasms, elevated PSA and urinary urgency. Ejaculatory dysfunction occurred in four patients in the Optilume arm and in 1 patient in the sham arm and no de novo erectile dysfunction was reported.

- Rezum Water Vapor Therapy: In recent years, the technology has been evaluated in a prospective, multicenter, double-blinded randomized controlled study conducted by McVary et al. (Clinicaltrials.gov: NCT01912339). Fifteen participating sites in the United States recruited 197 patients with moderate-to-severe LUTS with a prostate size from 30 cc to 80 cc. In this trial, 136 patients were assigned to the water vapor thermal therapy arm and 61 patients to the sham/control procedure. The primary efficacy endpoint was the change in the International Prostate Symptom Score (IPSS) from baseline to 3 months. Additionally, clinical events committees reviewed the safety of the device.

At the 3 months, the water vapor thermal therapy showed an IPSS reduction of 50% whereas the reduction was only 20% in the control group (p<0.0001). Moreover, other measurements such as Qmax, Qol (p<0.0001) and BHPII (p=0.0003) significantly improved in the Rezum therapy group when compared to the control group. Three serious adverse events (AE) occurred in two patients. One patient had de novo extended urinary retention and the second patient had nausea and vomiting. Moderate to severe AEs resolved within 3 weeks.

A 4-year outcomes of this trial was reported. Improvement of LUTS remain durable throughout 4 years with a reduction of 47% of the IPSS, 43% of the quality of life (QoL), and 52% of the Benign Prostatic Hyperplasia Impact Index. In addition, the retreatment rate was 4.4% at 4 years with no disturbances of sexual function.

C- Clinical investigation design

1. Objectives: The primary objective of the present study is to evaluate and compare patient experience, symptom relief and functional improvement when using Optilume® BPH Catheter System and RezumTM Water Vapor Therapy within 100 patients through several timepoints.
2. Sample size: OptiZum is a prospective, single center (Centre hospitalier Universitaire de Montréal), randomized, blinded clinical trial. The investigators expect to recruit 100 participants with a block randomization methodology to either Optilume® BPH Catheter System or RezumTM Water Vapor Therapy (50 participants in each arm).
3. Study duration: Enrollment is expected to take 12 months. Each participant will be followed post-operatively through 1 year with 1 week, 1 month, 3 months, 6 months and 12 months follow-up visits.
4. Number of sites: 1 site (Centre Hospitalier de l'Université de Montréal)
5. Point of enrollment: Each patient will be assigned a study ID after signing the informed consent form.

   * Investigators will be responsible for obtaining consent using the current study-specific, REB-approved consent documents prior to any baseline testing for eligibility that goes beyond standard care.
   * Participants will be consented in a manner understandable by the intended patient population and providing adequate time to address any questions or concerns.
   * Documentation of the consenting process and the signed/dated consent documents will be filed in the study Trial Master File.

   An informed consent form must be signed by each patient prior to study enrollment. Informed consent will be obtained according to the Declaration of Helsinki ("Ethical Principles for Medical Research Involving Human Subjects", The World Medical Association Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013), requirements of the standard ISO 14155:2020 ("Clinical investigation of medical devices for human subjects-Good clinical practice"), and individual institution guidelines.

   Re-consent will be required where changes are implemented, new information becomes available, or as required by regulations, and re-consent is needed.
6. Study visits and exams:

   6.1. Study visits:

   -Screening and baseline : Potential participants will undergo screening at the study center. Any study specific testing for eligibility determination that goes beyond standard care must be performed after REB approved study specific informed consent form is signed by the patients.

   Baseline tests and questionnaires will be completed 3 months maximum prior to the procedure.
   * Preoperative instructions : Patients will be instructed to stop anticoagulants and aspirin 3-5 days prior to the procedure depending on the type of anticoagulation.
   * Anesthesia : Optilume BPH Catheter System and Rezum water vapor therapy will be performed under general, spinal or local anesthesia .
   * Follow-ups : Participants will have 5 follow-up visits after the procedure. Patients will be seen in person for evaluation after 1 week, 1 month, 3 months, 6 months and 12 months following the procedure. Uroflowmetry will be performed and questionnaires will be completed by participants (IPSS, IIEF, MSHQ-EjD, Quality of recovery, Satisfaction).

   First follow-up visit will be performed 7 days +/- 5 days (1week follow-up visit). Second follow-up visit will be performed 28 days +/- 7 days (1 month follow-up visit). Third, fourth and fifth (3, 6 and 12 months follow-up visit) will be performed 90 days +/- 10 days , 180 days +/- 30 days and 360 days +/- 30 days).

   6.2. Study assessments :

   Several tests and questionnaires will be completed during this trial:
   * Uroflowmetry: participants will undergo measurement of urinary flow rate (Qmax), urinary mean flow rate (Qmean), total voided volume (TVV), and post-void residual volume (PVR). For an uroflowmetry test to be valid, the voided volume must be ≥ 125 mL. If the total voided volume is less than 125mL, the voided volume must be equal to or greater than 50% of the bladder capacity (defined as voided volume + PVR). The test can be repeated if necessary.
   * International Prostate Symptom Score (IPSS): IPSS is a validated measure of urinary symptoms due to BPH. The questionnaire will be completed at baseline and at follow-up visits.
   * International Index of Erectile Function (IIEF) (10): IIEF is a validated questionnaire used to assess erectile dysfunction. The questionnaire will be completed at baseline and at follow-ups visits.
   * Male Health Questionnaire for Ejaculatory Dysfunction (MSHQ-EjD) : MSHQ-EjD is a validated questionnaire used to assess ejaculatory function. The questionnaire will be completed at baseline and at follow-ups visits.
   * Transrectal ultrasound (TRUS): TRUS is performed to measure patient's prostate size at baseline.

   IPSS, QoL, IIEF, MSHQ-EjD, uroflowmetry and TRUS are standard of care tests and questionnaires.
   * Pain score: A visual Analog Scale (VAS) will be used to assess pain before and after the procedure.
   * Anxiety Symptoms Questionnaire (ASQ) (12): A questionnaire will be used to assess the intensity and frequency of symptoms related to anxiety.
   * Satisfaction: A questionnaire will be used to assess patient recovery at 1 month.

   D- Risk/benefit analysis

   - Optilume® BPH Catheter System: After treatment with the Optilume BPH Catheter System, the probable benefit is the relief of LUTS maintained at 1 year and the improvement of QoL, as showed by the PINNACLE study.

   The FDA summary of safety and effectiveness data (SSED) of the Optilume BPH Catheter System reported possible risks related to the use of the device. According to the report, potential AEs are similar to standard cystoscopic procedures and mechanical dilation. Potential AEs includes and are not limited to the following:
   * Fever
   * Bleeding
   * Pain
   * Urinary tract infection
   * False route of the urethra
   * Dysuria
   * Difficult urination
   * Frequency/urgency/irritative urinary symptoms
   * Urinary retention and related symptoms
   * Blood in urine (hematuria)
   * Urinary incontinence
   * Urethrorrhagia
   * Blood in semen (hematospermia)
   * Ejaculatory dysfunction
   * Bladder perforation
   * Urethral and/or bladder neck strictures
   * Injury or perforation to the urethra
   * Sphincter or prostatic capsule
   * Inflammation of genitourinary system (prostatitis, orchitis, balanitis)

   Additionally, some AEs can occur secondary to the use of paclitaxel coating. Systematic effects of this medication are not anticipated, however, intravenous paclitaxel used in chemotherapy is responsible of AEs. They include and are not limited to:
   * Allergic reaction
   * Alopecia
   * Anemia
   * Gastrointestinal symptoms
   * Hematological dyscrasia (including leucopenia, neutropenia, thrombocytopenia)
   * Hepatic enzyme changes
   * Myalgia/arthralgia
   * Myelosuppression
   * Peripheral neuropathy

     - RezumTM Water Vapor Therapy: According to Boston scientific, most patients will experience symptom relief in as soon as 2 weeks, with a maximum benefit at approximatively 3 months. Other potential benefits include:
   * Surgical retreatment rate: after 5 years, only 4.4% of patients needed another surgery for BPH symptoms
   * Does not typically require general anesthesia
   * No permanent implant
   * Preserves sexual function
   * Symptom relief that lasts

   However, potential risks include and are not limited to:
   * Painful or frequent urination
   * Blood in the urine or semen
   * Decrease in ejaculatory volume
   * Urinary tract infection (UTI)
   * Inability to urinate or completely empty the bladder
   * Urgent need to urinate
   * Inability to ejaculate
   * Urinary incontinence
   * Inflammation of the epididymis
   * Worsening erectile dysfunction
   * Pain/discomfort with ejaculation
   * Pelvic or penile pain/discomfort
   * Poor or splayed urine stream
   * Inflammation of the prostate gland
   * Scarring and narrowing of the urethra In rare occasion, the following AEs may occur including narrowing of the bladder neck, bladder stone, and severe infection. In addition, patient may experience continued of worsening BPH symptoms during healing phase.

   E- Ethical oversight:

   This study will be conducted in accord with the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans (2014), as well as in respect of the requirements set out in the applicable standard operation procedures of the Research Institute of the University of Montreal Health Care Center and of the University of Montreal Health Care Center Research Ethics Board. The University of Montreal Health Care Center Research Ethics Board will review this study and will be responsible for monitoring it.

   F- Data collection and storage: REDCap (a secure online software designed to manage surveys and e-consent forms) and Case report forms (CRFs) will be used to collect all subject data during the study. Data will be stored for 10 years as per institution requirements.

   G- Funding: The present study in funded by Laborie (Urotronic).

   H- Conflict of interest: Although this is an investigator-initiated study, it should be noted that the principal investigator (Dr Naeem Bhojani) is a consultant for Laborie/Urotronic.

ELIGIBILITY:
Inclusion Criteria:

* Male subject with symptomatic BPH.
* Prostate size 30-100g.
* Able to complete the study protocol.

Exclusion Criteria:

* Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with follow-up requirements
* Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate
* Any prior minimally invasive intervention (e.g., TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
* Confirmed or suspected malignancy of prostate or bladder
* Active urinary tract infection (UTI) confirmed by culture
* History of overt urinary incontinence requiring use of pads NOTE: Pad usage for post-micturition dribble is acceptable
* Presence of confounding diagnoses impacting lower urinary tract symptoms or bladder function (e.g., urethral strictures, bladder neck contracture, neurogenic bladder, detrusor instability, bladder stones, etc.)
* History of chronic urinary retention (e.g., PVR ≥300mL on two separate occasions, or catheter dependent drainage)
* Anatomy (e.g., presence of false passage or size of meatus) is not suitable for treatment with the Optilume BPH Catheter System
* Significant obstruction from median lobe (investigator opinion)
* Disease or other health condition that is not suitable for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The rate of patients without a catheter (catheter free) | 3 days
  The primary efficacy endpoint is defined as the rate of patients without a catheter (catheter free) 3 days after the procedure.
Frequency and severity of treatment related adverse events | Through study completion, an average of 2 years
  The primary safety endpoint is defined as the frequency and severity of treatment related adverse events reported using the Clavien-Dindo severity grading system.

OTHER OUTCOMES:
The change of the International Prostate Symptom Score (IPSS) | Baseline, 1week, 3, 6, 12 months.
  * The International Prostate Symptom Score (IPSS) change from baseline to 3, 6 and 12 months.
  * Score : 0-7 (Mild), 8 to 19 (Moderate), 20 to 35 (Severe)
International Prostate Symptom Score (IPSS) Quality of Life (QoL) | Baseline, 1week, 3, 6, 12 months.
  IPSS Quality of Life (QoL) change from baseline to 3, 6 and 12 months. Minimum value : 0 (Delighted) Maximum value : 6 (Terrible)
Maximum Flow Rate (Qmax) | Baseline, 1week, 3, 6, 12 months.
  Qmax change from baseline to 3, 6 and 12 months.
Post-Void Residual Volume (PVR) | Baseline, 1week, 3, 6, 12 months.
  PVR change from baseline to 3, 6 and 12 months.
International Index of Erectile Function (IIEF-5) | Baseline, 1week, 3, 6, 12 months.
  * IIEF change from baseline to 3, 6 and 12 months.
  * Score : 5-7 Severe Erection dysfunction; 8-11 Moderate Erection dysfunction; 12-16 Mild to Moderate Erection dysfunction;17-21 Mild Erection dysfunction
Male Sexual Health Questionnaire Ejaculatory Function (MSHQ-EjD) Short Form (MSHQ-EjD). | Baseline, 1week, 3, 6, 12 months.
  MSHQ-EjD change from baseline to 3, 6 and 12 months. Minimum value : 1 (Potential ejaculatory malfunction) Maximum value : 15 (Suggestive of normal ejaculation function)
Pain score (Visual Analog Scale). | 1 day
  * Pain score during/after the procedure (VAS)
  * Minimum value : 0 (No pain)
  * Maximum value : 10 (Pain as bad as it could possibly be)
Recovery time | 1 day
Quality of recovery-15 (QoR-15) | 30 days after the surgery
  Quality of recovery-15 (QoR-15) classification :
  * QoR-15 > 135 : Excellent
  * 122 ≤ QoR-15 ≤ 135 : Good
  * 90 ≤ QoR-15 ≤ 121 Moderate
  * QoR-15 < 90 : Poor
Number of calls to nurse/staff | 3 months
Number of returns to emergency room | 3 months
Patient satisfaction | 1 month, 3month
  Using a scale from 1 to 10, how satisfied are participants with their recovery and post-operative experience overall.
  Minimum : 1 (Being very dissatisfied) Maximum : 10 (Being very satisfied)
Patient anxiety | Baseline, 1 week
  The Anxiety Symptoms Questionnaire (ASQ) will be used to assess the intensity and frequency of symptoms related to anxiety. ASQ is scored on a scale of 0 to 340 with higher scores indicating greater anxiety severity. Intensity and frequency subtotals also range from 0 to 170.
  Minimum : 0 Maximum : 340
Surgical and medical retreatment rate | Through study completion, an average of 1 year
  Surgeries, use of alpha-blockers or 5alpha reductase inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Bhojani, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Dixon CM, Rijo Cedano E, Mynderse LA, Larson TR. Transurethral convective water vapor as a treatment for lower urinary tract symptomatology due to benign prostatic hyperplasia using the Rezum((R)) system: evaluation of acute ablative capabilities in the human prostate. Res Rep Urol. 2015 Jan 30;7:13-8. doi: 10.2147/RRU.S74040. eCollection 2015. PMID 25674555
- [Background] Baker A, Simon N, Keshaviah A, Farabaugh A, Deckersbach T, Worthington JJ, Hoge E, Fava M, Pollack MP. Anxiety Symptoms Questionnaire (ASQ): development and validation. Gen Psychiatr. 2019 Dec 18;32(6):e100144. doi: 10.1136/gpsych-2019-100144. eCollection 2019. PMID 31922090
- [Background] Rosen RC, Catania JA, Althof SE, Pollack LM, O'Leary M, Seftel AD, Coon DW. Development and validation of four-item version of Male Sexual Health Questionnaire to assess ejaculatory dysfunction. Urology. 2007 May;69(5):805-9. doi: 10.1016/j.urology.2007.02.036. PMID 17482908
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Background] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Background] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Background] Kaplan SA, Moss J, Freedman S, Coutinho K, Wu N, Efros M, Elterman D, D'Anna R, Padron O, Robertson KJ, Lawindy S, Mistry S, Shore N, Spier J, Kaminetsky J, Mazzarella B, Cahn D, Jalkut M, Te A. The PINNACLE Study: A Double-blind, Randomized, Sham-controlled Study Evaluating the Optilume BPH Catheter System for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2023 Sep;210(3):500-509. doi: 10.1097/JU.0000000000003568. Epub 2023 Aug 9. PMID 37555604
- [Background] Optilume® BPH Catheter System - FDA SUMMARY OF SAFETY AND EFFECTIVENESS DATA (SSED). FDA; 2023
- [Background] Santos Dias J. Benign prostatic hyperplasia: clinical manifestations and evaluation. Tech Vasc Interv Radiol. 2012 Dec;15(4):265-9. doi: 10.1053/j.tvir.2012.09.007. PMID 23244722
- [Background] Berry SJ, Coffey DS, Walsh PC, Ewing LL. The development of human benign prostatic hyperplasia with age. J Urol. 1984 Sep;132(3):474-9. doi: 10.1016/s0022-5347(17)49698-4. PMID 6206240